CLINICAL TRIAL: NCT05047757
Title: Fava Bean Protein and Amino Acid Bioavailability in Healthy Volunteers
Brief Title: Amino Acid Bioavilability of Fava Beans
Acronym: Leg4Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: University of Helsinki (Other); AgroParisTech (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, Professor, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Leg4LifeDIG
Record Dates: First submitted 2021-06-15; First posted 2021-09-17 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Ileal Digestibility of Amino Acids
Keywords: digestibility; healthy humans; nasoileal tubes; stable isotopes; legumes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fava bean (Experimental): The intervention consists in a test meal containing 250 g of cooked and peeled favabean, to provide 20 g protein. Fava bean are intrinsically labelled with 15N.
  Interventions: Dietary Supplement: Test meal with 15N labeled favabean

INTERVENTIONS:
Dietary Supplement: Test meal with 15N labeled favabean — Ingestion of a 15N labeled test meal. Subjects are equipped with a nasoileal tube. 15N is followed in biological fluids (plasma, effluents, urines).

SUMMARY:
The goal of the project is to determine the ileal amino acid digestibility of Favabean in healthy subjects equipped with naso-ileal tube. For this purpose, Favabean will be intrinsically labelled with 15N using 15N fertilizer. This procedure will be realized in Finland and the labelled material will be sent to the Unit PNCA.

DETAILED DESCRIPTION:
The objective is to determine the nutritional quality of protein from favabean in healthy humans, especially in terms of amino acid digestibility. Ileal digestibility is determined in ileal digesta collected postprandially with a naso-ileal tube. The favabeans are intrinsically labelled in 15N in order to track dietary nitrogen and amino acids in the samples.

Ethical and regulatory aspects:

The protocole was submitted to the Ethical Committee for approval and to the French Agency of Drugs and Health for administrative authorization. The personal data management will be in accordance with the regulation on personal data protection ( " regulation n° 2018-493 du 20 juin 2018").

Meal:

The meal will consist in 250 g of cooked and peeled favabean, to provide 20 g protein. Sensory tests will be realized to optimize the organoleptic properties of the meal. 15N labelled bean will be boiled in water with salt. On the morning of the experiment, the portion of fava bean will be warmed up.

Volunteers:

Eight subjects will be included in the study. The investigators plan to recruit around 16 volunteers to accommodate for the usual 50% dropouts.

One week before the experiment, the volunteers will follow a standard diet adapted to their body weight to control their protein intake (1.3 g protein/kg body weight). They will be ask to consume one to 3 portions of favabean in the week.

The volunteers will arrive at the Human Nutrition Research Centre of Avicenne Hospital on the morning before the day of the experiment. They will be equipped with a double lumen intestinal tube that will be allowed to progress through the intestinal tract for 24h. One of the lumen is radio opaque and serves to perfuse a non-absorbable maker in the intestine (slow marker method). The other lumen is dedicated to the continuous aspiration of the effluents, 15 cm below the perfusion site. The measurement of the non-absorbable marker in the effluents allows the determination of the effluent flow rate.

On the day of the experiment, the position of the tube will be checked by radiography to verify its location at the terminal ileum. A catheter will be inserted in the forearm vein for blood sampling. The perfusion of the non-absorbable marker, PEG-4000 (20g/l), will start at a flow rate of 1ml/min. The intestinal flow and the basal ileal sample will be collected during 30 min. Basal plasma sample will be sampled.

Then, at t=0, the volunteers will drink the test-meal. Until t=8h, intestinal content will be continuously collected by aspiration and pooled every 30 minutes. Blood will be sampled every 30 minutes during 4h and hourly thereafter. The urine will be collected every 2 h for 8 h.

Subjects will collect stools samples at home during the 48 h after the meal. Stools will be sent to Finland.

Measurements:

In the digesta:

PEG-4000 by turbidimetric method, total N and 15N enrichment by EA-IRMS, amino acid concentrations by UPLC (after acid hydrolysis HCl 6N at 110°C for 24h), 15N amino acid enrichment by GC-c-IRMS (after purification on cation exchange resin and derivatization).

In the plasma:

Glucose, urea (colorimetric methods), insulin (ELISA), amino acid concentrations (UPLC), 15N enrichment in plasma protein, urea and free amino acids (EA-IRMS, after purification on cation exchange resin and derivatization).

In the urine:

Urea (colorimetric method) and 15N urea (EA-IRMS, after purification on cation exchange resin and derivatization).

In the stools:

Micriobial DNA.

Outcomes:

Real ileal digestibility of protein and amino acids (digestive losses), Postprandial deamination (metabolic losses), Net Postprandial Protein Utilization, Microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* 18<BMI<30
* Good health (WHO=0)
* For woman: use of birth control

Exclusion Criteria:

* allergy against legumes
* allergy against latex
* pregnant women
* Positive serology for AgHBS, AcHbc, HCV, HIV
* Positive PCR test for SARS-Cov2
* Anemia
* Excessive alcohool consumption
* Hypertension, diabetes, digestive, hepatic or renal diseases, cardiac disease
* Exercice>7h/week
* Blood donation within 3 months before the study
* Participation to another clinical study within 3 months before the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Ileal digestibility of protein and amino acids | -30 minutes to 8 hours after the test meal
  The measurement of nitrogen (mmol) and 15N enrichment (atom %) in ileal samples allow to determine the amount of dietary nitrogen in the lumen. The measurement of amino acid concentration (mmol) and their individual 15N enrichment (atom %) allow the determination of dietary amino acids remaining in the lumen.
  Dietary amino acids and dietary nitrogen that are recovered in the ileal samples are then considered as non absorbed.

SECONDARY OUTCOMES:
Net Postprandial Protein Utilization (NPPU) | 0 to 8 hours after the test meal
  The measurement of urea (mmol) and 15N enrichment of urea (atom %) allow to determine the amount of dietary N that was transferred to urea, thus accounting for metabolic losses. Metabolic losses of dietary N, together with digestive losses of dietary N, are not retained in the body.
gut microbiota in response to the ingestion of 15N fava bean | 0 to 2 days after the test meal
  Microbial DNA sequencing
Nitrogen metabolites in blood in response to the ingestion of 15N fava bean | 0 to 8 hours after the test meal
  urea and amino acids (mmol/l)
Plasma glucose in blood in response to the ingestion of 15N fava bean | 0 to 8 hours after the test meal
  plasma glucose (mmol/l)
Plasma insulin in blood in response to the ingestion of 15N fava bean | 0 to 8 hours after the test meal
  plasma insulin (pmol/l)
Starch digestibility in response to the ingestion of fava bean | -30 minutes to 8 hours after the test meal
  The measurement of glucose from starch in ileal samples allow to determine the amount of undigested starch in the lumen.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Gaudichon, PhD, Prof, Study Director — AgroParisTech; Robert Benamouzig, MD, Prof, Principal Investigator — APHP
Locations (1):
- Centre de Recherche sur Volontaires (CRV), Hospital Avicenne, Bobigny, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Itkonen ST, Calvez J, Airinei G, Chapelais M, Khodorova N, Sahaka M, Benamouzig R, Stoddard FL, Simojoki A, Pajari AM, Gaudichon C. True Ileal Amino Acid Digestibility and Protein Quality of 15N-Labeled Faba Bean in Healthy Humans. J Nutr. 2024 Apr;154(4):1165-1174. doi: 10.1016/j.tjnut.2024.01.030. Epub 2024 Feb 3. PMID 38311065